CLINICAL TRIAL: NCT05336058
Title: A Case-control, Non-intervention Study for Gastric Cancer Screening
Brief Title: Development of Free DNA Multi-target Methylated PCR for Auxiliary Diagnosis of Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Singlera Genomics Inc. (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2201249-17
Record Dates: First submitted 2022-03-25; First posted 2022-04-20 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Stomach Cancer
Keywords: DNA methylation; Early gastric cancer screening
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric cancer group: We anticipate enrolling approximately 620 gastric cancer (GC) cases, comprising 20 sets of GC tumors and their corresponding peritumoral tissue samples, as well as a minimum of 600 plasma samples from patients across stages I to IV of GC. Pathological diagnosis is required.
  Interventions: Other: No intervention
- Negative group: A total of approximately 520 cases were included in the study, comprising 20 cases providing white blood cell samples from healthy individuals, and 500 patients diagnosed with gastric diseases other than gastric cancer (such as gastritis, atrophy, intestinal metaplasia, etc.), who provided plasma samples.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — In this non-intervention study, 10ml of whole blood of enrolled subjects was collected for multi-target PCR detection of cfDNA methylation.

SUMMARY:
This was a case control, non-intervention study jointly developed by Fudan University Cancer Hospital and Shanghai Singlera Genomics Company. The enrolled population was screened by gastric surgery, including gastric cancer, precancerous lesions, benign lesions, and healthy control group. 10ml of whole blood of the enrolled subjects was collected for multi-target PCR detection of cfDNA methylation. The objective is to explore the clinical performance of polygene methylation (PCR-fluorescence probe) in the adjunctive diagnosis of gastric cancer, including the sensitivity of detection of various types and stages of gastric cancer, the specificity of detection of healthy controls, precancerous states, precancerous lesions, and the detection interference of other cancers. The diagnostic performance will be compared with CA199, CEA and CA724. The research data will provide a basis for screening targets for the development of detection kits.

DETAILED DESCRIPTION:
Design and plan of the project: 1) Using the MONOD patent detection data of the company's previous research and combining with literature retrieval, analyze the tissue samples of gastric cancer of different stages and their paired paracancer tissues to screen the methylation mutation sites related to early gastric cancer and select the sites suitable for PCR detection; 2) ctDNA methylation markers in gastric cancer blood were preliminarily screened by plasma of healthy persons and preoperative plasma paired with tissues; 3) Using the screened blood ctDNA specific methylation markers, a targeted detection method for early gastric cancer lesions was designed; 4) The detection performance of the independent validation set sample confirmation establishment method.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age, no gender limitation;
2. those who can accept gastroscopy or provide pathological examination results of postoperative gastric biopsy
3. Patients newly diagnosed with stage I-IV gastric adenocarcinoma who had not received surgery, radiotherapy, chemotherapy, targeted therapy or other anti-tumor intervention before blood collection;
4. There were precancerous lesions and carcinoma in situ in the pathological examination of gastroscopy or esophageal biopsy, and no abnormalities in other gastric lesions, gastroscopy or other cancers. And no previous history of tumor disease.

Exclusion Criteria:

1. Previous digestive system tumors, including gastric cancer, esophageal cancer, colorectal cancer, liver cancer, etc.;
2. have a history of other cancers and have not been clinically cured (clinically cured: no recurrence and metastasis within 5 years after surgery);
3. Systemic inflammatory response syndrome;
4. A history of severe cardiovascular disease (e.g., previous myocardial infarction, coronary artery bypass grafting, or coronary stenting); A history of congestive heart failure; Patients with myocardial infarction within 6 months, uncontrolled severe hypertension, etc.) who were deemed unsuitable for inclusion by the investigator;
5. Those who have received major surgical treatment such as blood transfusion or transplantation within 3 months
6. Participants in other interventional clinical researchers, pregnant or lactating women, or patients with autoimmune diseases, genetic diseases, mental diseases, etc., within 3 months.
7. have participated in an "interventional" clinical trial within the past 30 days and have taken the experimental drug;
8. patients with other diseases deemed unsuitable for inclusion by the investigator;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants were recruited from the Department of Gastrosurgery, Fudan University Cancer Hospital, including gastric cancer, precancerous lesions of gastric cancer, other gastric lesions, no abnormalities in gastroscopy, and other cancers.
Sampling Method: Non-Probability Sample
Enrollment: 1140 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-04 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of methylation detection in gastric cancer | assessed up to 12 months
  To investigate the sensitivity and specificity of polygene methylation in the diagnosis of gastric cancer of different types and stages, and to evaluate its value as an auxiliary diagnosis.
Comparison of polygene methylation detection and other serological detection methods in gastric cancer | assessed up to 12 months
  The specificity and sensitivity of multigene methylation (PCR-fluorescence probe) and CA199, CEA and CA724 in the auxiliary diagnosis of gastric cancer were compared.
Screening of genetic targets for kit development | assessed up to 12 months
  The research data will provide a basis for screening gene targets for the development of subsequent detection kits.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Liu, PhD, Principal Investigator — Singlera Genomics Inc.
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu G, Wang GX, Wang HG, Mo FF, Tang BB. The value of detecting pepsinogen and gastrin-17 levels in serum for pre-cancerous lesion screening in gastric cancer. Neoplasma. 2019 Jul 23;66(4):637-640. doi: 10.4149/neo_2018_180825N647. Epub 2019 Apr 24. PMID 31058531
- [Background] Guo S, Diep D, Plongthongkum N, Fung HL, Zhang K, Zhang K. Identification of methylation haplotype blocks aids in deconvolution of heterogeneous tissue samples and tumor tissue-of-origin mapping from plasma DNA. Nat Genet. 2017 Apr;49(4):635-642. doi: 10.1038/ng.3805. Epub 2017 Mar 6. PMID 28263317
- [Background] Chen X, Gole J, Gore A, He Q, Lu M, Min J, Yuan Z, Yang X, Jiang Y, Zhang T, Suo C, Li X, Cheng L, Zhang Z, Niu H, Li Z, Xie Z, Shi H, Zhang X, Fan M, Wang X, Yang Y, Dang J, McConnell C, Zhang J, Wang J, Yu S, Ye W, Gao Y, Zhang K, Liu R, Jin L. Non-invasive early detection of cancer four years before conventional diagnosis using a blood test. Nat Commun. 2020 Jul 21;11(1):3475. doi: 10.1038/s41467-020-17316-z. PMID 32694610